CLINICAL TRIAL: NCT02117596
Title: Novel Pilot Trial of Sirolimus, Mycophenolate Mofetil, and Corticosteroids Versus a Historic Control Population Receiving Calcineurin Inhibitors Based Immunosuppression
Brief Title: Calcineurin Inhibitor Based Immunosuppression Withdrawal
Acronym: CNI-W
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pediatric Nephrology of Alabama (Other)
Collaborators: Pfizer (Industry); The Emmes Company, LLC (Industry)
Responsible Party: Principal Investigator, Mark Benfield, MD, MD, Pediatric Nephrology of Alabama
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CNI Withdrawal
Record Dates: First submitted 2014-04-16; First posted 2014-04-21 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-04

CONDITIONS: Renal Transplant
Keywords: Pediatric; Renal; Transplant
MeSH Terms: interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sirolimus (Other): Single arm
  Interventions: Drug: Sirolimus

INTERVENTIONS:
Drug: Sirolimus — 1. Tacrolimus (Prograf®) At 6 months post-transplantation, patients will have Prograf® tapered by 25% per week such that they will be off of this medication by 7 months post-transplantation.
  2. Sirolimus (Rapamune®):
  At 6 months post-transplantation, all patients will be administered Sirolimus at a dose of 1.65-2.79 mg/m2/day as a tablet or liquid (administered q 12 hours).
  Other Names: Rapamune; Rapamycin

SUMMARY:
Damage and scarring of a transplanted kidney has become the most common cause of loss of the transplanted kidney. This kidney damage is a complex process caused by many factors including injury during obtaining and transplanting the kidney, injury from the immune system, injury from infections, and injury from drugs used to stop rejection. This injury leads to scars that decrease the kidney's ability to function properly, and over time the kidney is lost. Prograf® (tacrolimus) has been one of the main drugs used to prevent rejection. However, when used over time it has been shown to cause chronic damage and scarring in the transplanted kidney.

The purpose of this experimental study is to determine whether children can safely be withdrawn from Prograf® after transplantation and changed to Rapamycin® (sirolimus). Recent research studies in adult transplantation have demonstrated that with the use of Rapamycin® (sirolimus), it is possible to discontinue the use of Prograf (tacrolimus) with no increase in rejection, with decreased scarring in the kidney, and with improvements in kidney function and survival of the kidney. A total of 50 children will enroll in this study at university centers around the country. This study will last about 3 years.

DETAILED DESCRIPTION:
Advances in immunosuppressive therapies in pediatrics have been associated with rapidly falling incidence of acute rejection and improving allograft survival. In recent analyses of the NAPRTCS database, acute rejection is no longer the most common cause of hospitalization or allograft failure. Chronic rejection has now become the most common cause of allograft failure and accounts for over 35% of allograft loss. Chronic rejection is a complex clinical condition that includes both immunologic and non-immunologic causes and is more accurately referred to as Chronic Allograft Nephropathy (CAN). Although Calcineurin inhibitors (CNI) have played a central role in reducing acute rejection and improving allograft survival, it has long been shown that they contribute to interstitial fibrosis and chronic allograft nephropathy. Recent trials in adult transplantation have demonstrated that with the use of the TOR-inhibitor, Sirolimus, it is possible to withdraw Calcineurin inhibitors with no increase in rejection and with improvements in allograft function, interstitial fibrosis and long term survival (1). We hypothesize that the use of Sirolimus (SRL) in pediatric kidney transplantation will allow the withdrawal of Calcineurin inhibitor and improved kidney function and long term survival. We plan to enroll 50 patients at the time of transplantation. Patients will receive routine immunosuppression of CNI (Prograf), Mycophenolate mofetil (Cellcept) and prednisone. Those patients with normal function and no rejection episodes after 6 months of transplantation will undergo a slow conversion from Prograf to Sirolimus (Rapamune). We will then assess the rate of rejection, allograft function, fibrosis on biopsy, and allograft survival over the following 18 months.

ELIGIBILITY:
Inclusion Criteria at Transplant:

* Age < 19 years (up to the day of the 19th birthday)
* Panel Reactive Antibody Level (PRA) <20% (Flow cytometry method)
* Recipient of first living donor or deceased donor renal transplantation
* Signed and dated informed consent (per local IRB standards)

Exclusion Criteria at Transplant:

* Recipients of multi-organ transplants (e.g. kidney/pancreas transplant, etc.)
* Peak PRA > 20% at any time
* Recipient of en-bloc kidneys
* Recipient of an organ from an HLA identical donor or a non-heart beating donor
* Pregnant or lactating
* Positive for HIV or an immunodeficiency virus
* History of malignancy
* Use of investigational agents within 4 weeks prior to transplantation
* Current use of terfenadine, cisapride, astemizole, or pimozide (unless discontinued before administration of SRL)
* Known hypersensitivity to sirolimus
* Known hypersensitivity to Prograf, Cellcept, prednisone, Cremophor, HCO-60, or murine products

Max Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 52 (Actual)
Dates: Start 2007-11; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
This study has a primary endpoint of allograft function as determined by Schwartz GFR at 18 months after conversion to CNI free protocol (2 years post transplantation). | 18 mos after conversion to CNI free protocol

SECONDARY OUTCOMES:
Secondary outcomes will include biopsy proven acute rejection episodes, progression of quantitative interstitial fibrosis as determined by Sirius Red staining and digital image analysis, Allograft survival and patient survival | measured at 12 and 24 months post transplant

CONTACTS AND LOCATIONS:
Overall Officials: Mark Benfield, M.D., Principal Investigator — Pediatric Nephrology of Alabama
Locations (4):
- United States (4):
  - Pediatric Nephrology of Alabama, Birmingham, Alabama
  - UCLA, Los Angeles, California
  - Stanford University, Stanford, California
  - Emory University, Atlanta, Georgia